CLINICAL TRIAL: NCT03750864
Title: An Innovative Approach to Reduce Lung Cancer Stigma
Brief Title: Innovative Approach to Reduce Lung Cancer Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 29927
Record Dates: First submitted 2018-11-09; First posted 2018-11-23 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer Stigma; Lung Cancer; Stigma, Social; Stigmatization; Acceptance Processes
Keywords: Lung cancer; Stigma; Lung cancer stigma; Acceptance and commitment therapy
MeSH Terms: conditions — Lung Neoplasms; Social Stigma; Stereotyping; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-LCS Therapy (Experimental): Intervention is psychosocial counseling utilizing Acceptance and Commitment Therapy for Lung Cancer Stigma (ACT-LCS) as a patient-focused intervention to reduce the self-blame, guilt and inhibited disclosure associated with lung cancer stigma.
  Interventions: Behavioral: ACT-LCS Therapy

INTERVENTIONS:
Behavioral: ACT-LCS Therapy — All participants in Stage 1, and those randomized to the intervention condition in Stage 2, will receive the Acceptance & Commitment Therapy for Lung Cancer Stigma (ACT-LCS) intervention. The ACT-LC intervention is designed to be delivered as 6 sessions of individual psychotherapy with a trained psychotherapist at a weekly or bimonthly rate, delivered either in person or over the phone. The treatment manual is based in Acceptance and Commitment Therapy (ACT). Therapists are instructed to begin treatment with Module 1. Modules 2-5 can then be administered in any order at the discretion of the therapist, based upon what the therapist thinks is most likely to be helpful to the patient. Module 6 is the final session of treatment.

SUMMARY:
This is a feasibility study examining the feasibility and acceptability of a novel psychotherapy intervention on lung cancer patients who are experiencing stigma.

DETAILED DESCRIPTION:
Experiences of stigma (perception and internalization of negative appraisal and devaluation from others) are pervasive for lung cancer patients. Previous work has shown associations between lung cancer stigma and detriments in clinically relevant outcomes such as depression, lower quality of life, and reduced engagement in cancer care.

The investigators previously developed Acceptance and Commitment Therapy for Lung Cancer Stigma (ACT-LCS) as a patient-focused intervention to reduce the self-blame, guilt and inhibited disclosure associated with lung cancer stigma. ACT-LCS is based in Acceptance and Commitment Therapy (ACT), a cognitive-behavioral treatment that promotes psychological flexibility through acceptance and valued direction.

This is a feasibility study examining the feasibility and acceptability of ACT-LCS.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in English
* Diagnosed with or treated for Non-Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer (SCLC) within the prior 12 months.
* Scores of 37.5 on the Lung Cancer Stigma Inventory (LCSI) screening measure

Exclusion Criteria:

* Not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Number of individuals who consent to the intervention | 10 months
  This measure will be calculated as a function of those eligible and approached who consented to the intervention. It will be utilized as a metric of feasibility and acceptability.
Number of sessions that each consented patient attended | 10 months
  This measure will be calculated as a count of sessions that each consented participant attended. It will be utilized as a metric of acceptability of the intervention among consented participants.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Hamann, PhD, Principal Investigator — University of Arizona; Linda Garland, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No